CLINICAL TRIAL: NCT00336830
Title: Improving Cardiac Rehabilitation Participation in Women and Men
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Neville Suskin, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: R-02-037; CIHR 56926 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Myocardial Infarction; Unstable Angina; Coronary Disease
Keywords: Cardiac Rehabilitation; Improving Cardiac Rehabilitation Participation; coronary angioplasty; coronary artery bypass surgery
MeSH Terms: conditions — Myocardial Infarction; Angina, Unstable; Coronary Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Active Comparator): Comparator without MD endorsement of Cardiac Rehabilitation
  Interventions: Behavioral: Standard Cardiac Rehabilitation referral
- MD Endorsment of CR (Experimental): Provided with MD endorsement of participation in Cardiac Rehabilitation
  Interventions: Behavioral: MD-endorsed Cardiac Rehabilitation referral

INTERVENTIONS:
Behavioral: MD-endorsed Cardiac Rehabilitation referral — Note to patient with general description of the Cardiac Rehabilitation program with signature and strong recommendation from attending physician.
  Other Names: MD endorsed referral to Cardiac Rehabilitation
  Arms: MD Endorsment of CR
Behavioral: Standard Cardiac Rehabilitation referral — Note to patient with general description of the Cardiac Rehabilitation program without signature or recommendation from attending physician.
  Other Names: Standard Referral to Cardiac Rehabilitation
  Arms: Usual Care

SUMMARY:
The purpose of this study is to determine the effect of a pre-discharge written personal endorsement to the patient by the patient's attending cardiologist or cardiac surgeon (MD endorsement) to take part in the Cardiac Rehabilitation and Secondary Prevention (CR) program, in addition to the standard CR referral, compared to the standard CR referral alone, on CR program enrollment within 2 months of index hospital discharge following admission for myocardial infarction, unstable angina, coronary angioplasty, or coronary artery bypass.

DETAILED DESCRIPTION:
There is compelling evidence that a comprehensive CR program comprising the delivery of lifestyle modifying education will reduce mortality, morbidity and improve quality of life in patients following myocardial infarction, angioplasty or, coronary artery bypass. However, less than 20% of eligible patients participate in CR programs. This study will look at a method of potentially improving enrollment and adherence to a CR program. It is expected that patients who receive the MD-endorsed referral will be more likely to attend the initial Orientation appointment and more closely adhere to the 6-month comprehensive CR program, as compared to the patients who receive a standard CR referral alone.

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to hospital for myocardial infarction (MI), unstable angina (UA), percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass surgery (CABS)
* Patient resides within 1 hour driving time from London

Exclusion Criteria:

* Inability to provide written informed consent or complete survey due to language or cognitive difficulties
* Previous cardiac rehabilitation participation
* Patient scheduled to undergo PTCA or CABS within two months following the index hospital discharge
* Inability to exercise due to musculoskeletal problems or previous or current stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2003-05; Primary Completion 2007-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Attendance at initial CR orientation appointment within 2 months of index hospital discharge | 3 months

SECONDARY OUTCOMES:
Impact of MD endorsement on number of patients attending CR program | 3 months
Number of patients who continue to adhere to the 6-month CR program beyond the initial CR orientation appointment | 8 months
Impact of other patient variables and how they influence participation in a CR program | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Neville Suskin, MBChB, MSc, Principal Investigator — University of Western Ontario & London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada